CLINICAL TRIAL: NCT07057401
Title: Investigation of Clinical Wear and Surface Roughness of Partial Restorations Fabricated Using Additive and Subtractive Manufacturing Methods: A Split-Mouth Randomized Controlled Clinical Trial
Brief Title: Evaluation of Clinical Wear and Surface Roughness of Partial Restorations Produced by Additive and Subtractive Manufacturing Methods: A Split-Mouth Randomized Controlled Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Husna Selinay (Other)
Responsible Party: Sponsor-Investigator, Husna Selinay, Research Assistant Dentist, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Department of Restorative Dent
Record Dates: First submitted 2025-06-03; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: CAD/CAM Space Maintainer; 3D Printing; Dental Treatment; Dental Disease
Keywords: subtractive manufacturing, additive manufacturing, roughness, wear
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: Evaluation of Wear and Surface Roughness of Partial Crowns Produced by Additive and Subtractive Manufacturing: A 1-Year Randomized Controlled Clinical Trial
Who Masked: Participant, Investigator
Masking Description: The aim of the study is to evaluate the wear values and surface roughness of single crown restorations performed on permanent molar teeth produced by CAD-CAM and 3D printing methods over a 12-month period using the Geomagic 3X device for wear measurement and a profilometer for roughness assessment.
  Participants will be systemically healthy individuals aged 18 to 50 years, with no periodontal support loss, indicated for crown restoration, and having natural antagonist teeth, who apply to the Department of Restorative Dentistry Clinic at Çukurova University Faculty of Dentistry.
  A total of 15 single crown restorations will be performed on first molar teeth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD-CAM Group (Experimental): Participants will receive single crown restorations manufactured by subtractive manufacturing (CAD-CAM milling) techniques.
  Interventions: Device: CAD-CAM Manufactured Crowns
- 3D Printing Group (Experimental): Participants will receive single crown restorations manufactured by additive manufacturing (3D printing) techniques.
  Interventions: Device: 3D Printed Crowns

INTERVENTIONS:
Device: CAD-CAM Manufactured Crowns — Single crowns produced using computer-aided design and milling technology applied to permanent molars.
  Arms: CAD-CAM Group
Device: 3D Printed Crowns — Single crowns produced using 3D printing technology applied to permanent molars.
  Arms: 3D Printing Group

SUMMARY:
The aim of this study is to compare the surface roughness and wear values of crowns fabricated using currently utilized 3D printing and CAD-CAM technologies.

In recent years, crown restorations produced with CAD-CAM systems have been safely used in dentistry. These types of restorative materials are expected not to undergo significant wear themselves and also not to cause wear on natural teeth. Therefore, the structural resistance and hardness of the material are clinically very important. Restorations produced using 3D printing are among the latest technological developments in dentistry.

Additive manufacturing has been defined by the American Society for Testing and Materials (ASTM) as "the process of joining materials layer upon layer to make objects from 3D model data, as opposed to subtractive manufacturing methodologies."

3D printers have started to be used in various disciplines of dentistry such as dental education, oral surgery, dental implantology, orthodontics, pedodontics, prosthodontics, and restorative dentistry. In restorative clinics, they can especially be used in intracoronal restorations. However, studies in this area are quite limited.

The objective of this study is to evaluate the wear values using a Geomagic 3X device and the surface roughness values using a profilometer device over a 12-month period on single crown restorations applied to permanent first molars fabricated by CAD-CAM and 3D printing techniques.

A total of 26 single crown restorations will be performed on first molars. Participants will be selected among individuals aged 18-50 who apply to the Department of Restorative Dentistry, Faculty of Dentistry, Çukurova University. Eligible individuals must be systemically healthy, have no periodontal attachment loss, have an indication for crown restoration, and have a natural opposing tooth in contact with the restored tooth.

DETAILED DESCRIPTION:
In today's dentistry, where aesthetics has gained increasing importance, the use of CAD-CAM in the fabrication of fixed prostheses has become widespread.

Although restorations produced by traditional methods are of high quality, they are mechanically and aesthetically affected due to being shaped manually by the dentist (conventional method). Therefore, errors that may occur during fabrication can negatively affect the durability and marginal adaptation of composite restorations.

In a study comparing production techniques, composite crowns produced by the direct technique and single crown restorations fabricated using CAD-CAM were examined under an electron microscope. The composite restorations manufactured with the indirect technique showed more porosity, while no porosity was observed in restorations produced with the CAD-CAM method.

This result may be attributed to the fact that the prefabricated CAD-CAM blocks are homogeneous and subjected to quality control during production. As a result, internal structural defects are generally not observed in milled products. The absence of porosity is an important factor in the durability and fit of restorations.

3D Printers Restorations produced using 3D printers are among the latest technological advancements in dentistry. Additive manufacturing has been defined by the American Society for Testing and Materials (ASTM) as "the process of joining materials layer upon layer to create objects from 3D model data, as opposed to subtractive manufacturing methodologies." 3D printers have begun to be used in various dental disciplines such as dental education, oral surgery, dental implantology, orthodontics, pedodontics, prosthodontics, and restorative dentistry. In restorative clinics, they can especially be utilized for intracoronal restorations. However, studies in this area remain quite limited.

Null hypothesis of this study is that there is no statistically significant difference in clinical wear and surface roughness between single crown indirect restorations fabricated using additive and subtractive manufacturing methods.

ELIGIBILITY:
Inclusion Criteria:

* Teeth with Devital and Vital Cusp Loss

Exclusion Criteria:

* Root Canal Treated Teeth with Lesions
* Symptomatic Vital Teeth

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-07-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Wear | 12 months
  Measuring wear value using the Geomagic 3X device
Surface roughness | 12 months
  Measuring surface roughness values using a profilometer device

CONTACTS AND LOCATIONS:
Overall Officials: ezgi sonkaya akburak, doctor lecturer, Study Director — Cukurova University Restorative Dentistry
Locations (1):
- Çukurova Üniversitesi, Adana, sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39900133/